CLINICAL TRIAL: NCT06962462
Title: Effect of Daily Tadalafil Therapy on Endothelin-1 and E-Selectin in Diabetic Patients With Erectile Dysfunction
Brief Title: Daily Tadalafil in Diabetic ED Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Khalid Abdelmawgoud, Resident Doctor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-AKA-001
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Erectile Dysfunction Associated With Type 2 Diabetes Mellitus
Keywords: Tadalafil, Endothelin-1, E-selectin, Diabetic complications, Sexual dysfunction, ELISA
MeSH Terms: conditions — Diabetes Complications; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tadalafil Group (Experimental): Diabetic male patients with erectile dysfunction will receive oral tadalafil 5 mg once daily for 3 months to assess changes in serum Endothelin-1 and E-selectin levels.
  Interventions: Drug: Methyl Cellulose Placebo
- Placebo Group (Placebo Comparator): Healthy male participants matched by age will receive oral placebo tablets (methyl cellulose) once daily for 3 months. Blood samples will be collected pre- and post-intervention for biomarker assessment.
  Interventions: Drug: Methyl Cellulose Placebo

INTERVENTIONS:
Drug: Methyl Cellulose Placebo — Oral administration of inert methyl cellulose placebo tablets once daily for 3 months. Used as a comparator in healthy control participants to evaluate changes in Endothelin-1 and E-selectin serum levels.

SUMMARY:
This study evaluates the effect of 5 mg daily tadalafil therapy on serum levels of Endothelin-1 and E-selectin in diabetic male patients with erectile dysfunction. Outcomes will be compared pre- and post-treatment versus healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Male patients aged between 30 and 60 yearsز Diagnosed with diabetes mellitus Suffering from erectile dysfunction No history of hypertension or other systemic diseases

Exclusion Criteria:

History of pelvic trauma or major pelvic surgery Pacientes con hipogonadismo o hiperprolactinemia Chronic liver disease or cardiovascular disorders Chronic use of central nervous system drugs, anti-androgenic drugs, or Tramadol Smokers Non-vasculogenic erectile dysfunction Known allergy to tadalafil

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Effect of tadalafil 5 mg on serum levels of Endothelin-1 and E-selectin | 3 months after intervention
  Measurement of serum Endothelin-1 and E-selectin concentrations in diabetic patients with erectile dysfunction, before and after daily tadalafil 5 mg for 3 months, using ELISA technique.

SECONDARY OUTCOMES:
Biochemical assessment of serum Endothelin-1 and E-selectin levels | 3 months after intervention
  Measurement of serum levels of Endothelin-1 and E-selectin in diabetic patients with erectile dysfunction using ELISA technique before and after tadalafil 5 mg daily treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelmawgoud, M.Sc, Principal Investigator — Faculty of Medicine, South Valley University

IPD SHARING:
Plan to Share IPD: No